CLINICAL TRIAL: NCT06890585
Title: A Randomized, Multicenter, Open-Label Phase II Clinical Study Comparing the Efficacy and Safety of Zanubrutinib, Chidamide, and Rituximab Induction Therapy Sequentially Combined With or Without CHOP Versus R-CHOP in the First-Line Treatment of Patients With Newly Diagnosed Double-Expressor Diffuse Large B-cell Lymphoma
Brief Title: Zanubrutinib, Chidamide, and Rituximab Induction With or Without CHOP Versus R-CHOP in Newly Diagnosed Double-Expressor DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Zhiming (Other)
Responsible Party: Sponsor-Investigator, Li Zhiming, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-849-01
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: BTK Inhibitors; Histone Deacetylase Inhibitor; Double Express Diffuse Large B-cell Lymphoma
Keywords: Double Expressor Diffuse Large B-cell Lymphoma; zanubrutinib; chidamide
MeSH Terms: interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZCR-CHOP (Experimental): Cycle 1-2 Drug: Zanubrutinib Zanubrutinib will be given at a dose of 160mg，bid，from d1 to d21 in a 21-day cycle Drug: Chidamide Chidamide will be given at a dose of 20 mg after breakfast on day 1, day 4, day 8, day 11 in a 21-day cycle Drug: Rituximab Rituximab will be given at a dose of 375 mg/m2 by IV on day 1 in a 21-day cycle
  Cycle 3-8 Patients who achieve complete response evaluated by PEC-CT per Lugano 2014 criteria after two course of treatment will continue to take Zanubrutinib, chidamide, and rituximab for up to 8 cycles in total.
  Patients who achieve partial response and stable disease will take ZCR combined with CHOP or up to 8 cycles in total.
  CHOP : cyclophosphamide 750 mg/m2 IV D1, Doxorubicin/Epirubicin 50 mg/m2 IV, vincristine 1.4 mg/m2 IV [maximum total 2 mg], and prednisone 30 mg orally tid from d1 to d5 in a 21-day cycle
  Interventions: Drug: ZCR-CHOP
- R-CHOP (Active Comparator): R-CHOP Rituximab 375 mg/m2 IV on d1, cyclophosphamide 750 mg/m2 IV on d1, Doxorubicin/Epirubicin 50 mg/m2 IV on d1, vincristine 1.4 mg/m2 IV [maximum total 2 mg] on d1, and prednisone 30 mg orally tid from d1 to d5 in a 21-day cycle for up to 6 cycles.
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: ZCR-CHOP — Zanubrutinib, Chidamide, and Rituximab Induction Therapy Sequentially Combined With or Without CHOP
  Arms: ZCR-CHOP
Drug: R-CHOP — R-CHOP
  Arms: R-CHOP

SUMMARY:
Zanubrutinib, as a new generation of BTK inhibitors, has shown more potent antitumor activity and lower adverse reactions than ibrutinib in head-to-head clinical studies, which make it a promising regimen for B cell lymphoma. Chidamide is an oral subtype-selective histone deacetylase inhibitor.

This Randomized, Multicenter, Open-Label Phase II Clinical Study is comparing the efficacy and safety of Zanubrutinib, Chidamide, and Rituximab induction therapy sequentially combined with or without CHOP versus R-CHOP in the first-line treatment of patients with newly diagnosed double-expressor DLBCL.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy and safety of zanubrutinib, chidamide, and rituximab (ZCR) induction therapy sequentially combined with or without CHOP regimen versus the standard R-CHOP regimen as first-line treatment for newly diagnosed double-expressor DLBCL. This study targets patients with MYC/BCL2 double-expressing DLBCL, a group with poor prognosis under traditional R-CHOP treatment.

The study consists of screening period, treatment period, and follow-up period, with subjects randomly assigned to the experimental group and the control group in a 1:1 ratio. The primary endpoint is the end-of-treatment complete response rate (EOT-CRR), while secondary endpoints include the overall response rate (EOT-ORR), duration of response (DOR), progression-free survival (PFS), overall survival (OS), and safety. A total of 128 patients are planned to be enrolled.

Efficacy evaluation will be conducted using the 2014 Lugano criteria, with imaging examinations such as PET-CT to objectively measure treatment response. adverse events (AEs) throughout the entire trial and grade the severity of adverse events will be recorded according to the guidelines of the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed MYC/BCL2 double-expressor DLBCL confirmed by pathological histology/clinical imaging, with IHC BCL2 expression ≥50% and MYC expression ≥40%.
* Male or female patients aged 18-65 years.
* ECOG score of 0-2.
* Expected survival time of ≥6 months.
* Must have at least one evaluable or measurable lesion according to the Lugano 2014 criteria [Evaluable lesion: lymph node or extranodal local uptake increased (higher than the liver) on 18F-Fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) scan, and PET and/or Computed Tomography (CT) features consistent with lymphoma; Measurable lesion: nodal lesion with a long diameter >15mm or extranodal lesion with a long diameter >10mm, with increased 18FDG uptake]. Patients with no measurable lesions and diffuse 18FDG uptake in the liver should be excluded.
* Good major organ function, meeting the following requirements within one week before enrollment: blood routine WBC ≥3×10^9/L, Hb ≥80g/L, PLT ≥80×10^9/L; normal cardiac and liver function (total bilirubin ≤1.5 times the upper limit of normal, ALT and AST ≤2.5 times the upper limit of normal), normal renal function (serum creatinine ≤1.5 times the upper limit of normal), and no coagulation abnormalities.
* LVEF ≥50% as measured by echocardiography.
* Women of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment and be willing to use reliable contraception during the study.
* Subjects voluntarily join the study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Special types of DLBCL:Fluid overload-associated large B-cell lymphoma, primary mediastinal large B-cell lymphoma, mediastinal gray zone lymphoma, primary central nervous system (CNS) DLBCL, double-hit DLBCL with BCL2 and MYC rearrangements.
* Transformed DLBCL (e.g., DLBCL transformed from follicular lymphoma, chronic lymphocytic leukemia/small B-cell lymphoma), secondary CNS involvement of DLBCL.
* History of other malignancies within the past 5 years, except for squamous cell carcinoma of the skin, basal cell carcinoma of the skin, and carcinoma in situ of the cervix.
* Major surgery within the past 2 months (excluding diagnostic surgery).
* Previous treatment for NHL, including chemotherapy, immunotherapy, radiotherapy, monoclonal antibody therapy, or surgical treatment (excluding diagnostic surgery and biopsy).
* Previous treatment with cytotoxic drugs or anti-CD20 monoclonal antibody therapy for other diseases (e.g., rheumatoid arthritis).
* Use of any monoclonal antibody within 3 months prior to enrollment, participation in other clinical trials with investigational drugs, or vaccination with live attenuated virus vaccines within 1 month prior to enrollment.
* Use of hematopoietic growth factors within 2 weeks prior to enrollment.
* Suspected active or latent tuberculosis.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infections (excluding nail bed fungal infections) within 4 weeks prior to enrollment, or any major systemic infection requiring intravenous antibiotics or hospitalization (excluding tumor fever).
* History of severe bleeding disorders, such as hemophilia A, hemophilia B, von Willebrand disease, or spontaneous bleeding requiring transfusion or other medical intervention.
* HIV-positive patients. Active HBV-positive and HCV-positive patients, but those with controlled conditions as judged by the investigator may be cautiously enrolled with effective antiviral intervention.
* Other severe diseases that may limit participation in this trial, such as uncontrolled diabetes; severe heart failure (NYHA class II or above); acute coronary syndrome within the past 6 months; coronary revascularization within the past 6 months, such as stent implantation, coronary artery bypass grafting, and other heart and large vessel surgeries; severe arrhythmias including frequent premature ventricular contractions, ventricular tachycardia, rapid atrial fibrillation/flutter, severe bradycardia. Uncontrolled hypertension (greater than 150/100 mmHg). Gastric ulcer (with a risk of perforation as judged by the investigator); active autoimmune diseases; severe hypertension; severe respiratory diseases (e.g., obstructive pulmonary disease and bronchospasm history), such as known interstitial pneumonia or highly suspected interstitial pneumonia; or patients who may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Contraindications to any study drug, including previous treatment with anthracyclines; patients with diabetes who cannot tolerate prednisone treatment in this regimen.
* History of alcohol abuse or drug abuse.
* Allergic constitution, or known allergy to any active ingredient, excipient, or murine products, heterologous proteins included in this study.
* Requirement for continuous treatment with strong CYP3A inhibitors or inducers (see Appendix 6).
* Severe mental illness.
* Patients unable to comply with the study and/or follow-up phases.
* Patients unable to swallow study drugs normally.
* Patients deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
EOT-CR | Approximately 12 months
  defined as the proportion of subjects with measurable disease who achieve CR at the end of treatment according to 2014 Lugano criteria

SECONDARY OUTCOMES:
EOT-ORR | Approximately 12 months
  defined as the proportion of subjects with measurable disease who achieve CR and PR at the end of treatment according to 2014 Lugano criteria
Duration of response（DOR） | Approximately 24 months
  defined as the time from the date of first occurrence of CR or PR to the date of the first documented PD or death due to any cause according to 2014 Lugano criteria.
Progression-free survival (PFS) | Approximately 24 months
  defined as the time from treatment to disease progression or death from any cause according to 2014 Lugano criteria.
Overall survival (OS) | Approximately 24 months
  defined as the time from treatment to death from any cause according to 2014 Lugano criteria.
Adverse Events (AE) | Approximately 12 months
  all adverse events occurring during or after the first treatment will be summarized by treatment arm and NCI CTCAE grade.

OTHER OUTCOMES:
The consistency between ctDNA clearance and radiographic disease response | Approximately 12 months
  ctDNA will be collected from patients in the experimental group at baseline, the end of cycle 2, and the end of treatment. This includes, but is not limited to, evaluating the relationship between the clearance of the MYD88 L265P mutation and radiographic complete response after cycle 2 and at the end of treatment, as well as the relationship between the clearance of TP53 mutations and radiographic complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No